CLINICAL TRIAL: NCT02893293
Title: Imaging of Osteonecrosis With Ferumoxytol-Enhanced MRI
Acronym: Osteonecro
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Heike E Daldrup-Link, Professor of Radiology, Stanford University
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB-20253(osteonecrosis); PEDSBONE0006 (Other: OnCore)
Record Dates: First submitted 2016-07-27; First posted 2016-09-08 (Estimated); Results first posted 2024-11-26 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-10

CONDITIONS: Osteonecrosis
MeSH Terms: conditions — Osteonecrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ferumoxytol-enhanced MRI (Active Comparator): Patients receive a ferumoxytol injection (Feraheme, AMAG, 5mg Fe/kg, single administration) prior to routine decompression surgery and autologous stem cell transplant. Follow-up imaging with magnetic resonance imaging will be conducted in regular intervals for evaluation of the response to treatment.
  Interventions: Drug: Ferumoxytol-enhanced magnetic resonance imaging; Device: Magentic Resonance Imaging
- Non-ferumoxytol enhanced MRI (Sham Comparator): Patients scheduled for routine decompression surgery and autologous stem cell transplant will receive follow-up magnetic resonance imaging in regular intervals for evaluation of the response to treatment.
  Interventions: Device: Magentic Resonance Imaging

INTERVENTIONS:
Drug: Ferumoxytol-enhanced magnetic resonance imaging — Eligible patients receive a single ferumoxytol-dose and follow-up magnetic resonance imaging to evaluate success of stem cell transplant
  Arms: Ferumoxytol-enhanced MRI
Device: Magentic Resonance Imaging — Both arms will receive MRI
  Other Names: MRI

SUMMARY:
The goal of the project is to evaluate osteonecrosis before and after decompression surgery with ferumoxytol-enhanced MRI.

DETAILED DESCRIPTION:
The goal of the project is to evaluate osteonecrosis before and after decompression surgery with ferumoxytol-enhanced MRI.

The investigators approach relies on the FDA-approved iron supplement ferumoxytol (Feraheme), which is used off label as a contrast agent for MRI. Ferumoxytol is composed of iron oxide nanoparticles, which provide a strong T1- and T2-signal on magnetic resonance (MR) images and are taken up by cells in bone marrow.

20 patients will undergo MRI before and after decompression surgery and transplantation of bone marrow derived cells. 10 patients will receive a single intravenous injection of ferumoxytol prior to their surgery. 10 additional patients will serve as untreated controls. The investigators hypothesize that MR images after intravenous injection of ferumoxytol will improve lesion detection and allow to track transplanted bone marrow cells. MR imaging findings will be correlated with clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Osteonecrosis
* planned decompression surgery with autologous stem cell transplant

Exclusion Criteria:

* Contraindications for magnetic resonance imaging
* Hemosiderosis/hemochromatosis ( patients can still be included in the non-ferumoxytol arm)

Ages: 8 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 14 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heike Daldrup-Link, MD, PhD, Principal Investigator — Stanford University
Locations (1):
- Lucile Packard Children's Hospital, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Muehe AM, Feng D, von Eyben R, Luna-Fineman S, Link MP, Muthig T, Huddleston AE, Neuwelt EA, Daldrup-Link HE. Safety Report of Ferumoxytol for Magnetic Resonance Imaging in Children and Young Adults. Invest Radiol. 2016 Apr;51(4):221-227. doi: 10.1097/RLI.0000000000000230. PMID 26656202
- [Background] Nejadnik H, Lenkov O, Gassert F, Fretwell D, Lam I, Daldrup-Link HE. Macrophage phagocytosis alters the MRI signal of ferumoxytol-labeled mesenchymal stromal cells in cartilage defects. Sci Rep. 2016 May 13;6:25897. doi: 10.1038/srep25897. PMID 27174199
- [Result] Theruvath AJ, Nejadnik H, Muehe AM, Gassert F, Lacayo NJ, Goodman SB, Daldrup-Link HE. Tracking Cell Transplants in Femoral Osteonecrosis with Magnetic Resonance Imaging: A Proof-of-Concept Study in Patients. Clin Cancer Res. 2018 Dec 15;24(24):6223-6229. doi: 10.1158/1078-0432.CCR-18-1687. Epub 2018 Sep 17. PMID 30224340
- See also: Pediatric Molecular Imaging Program — http://daldrup-link-lab.stanford.edu/

RESULTS

PARTICIPANT FLOW:
Groups:
- Ferumoxytol-enhanced MRI: Patients scheduled for routine decompression surgery and autologous stem cell transplant receive ferumoxytol injection (Feraheme, AMAG, 5mg Fe/kg, single administration), and follow-up magnetic resonance imaging in regular intervals for evaluation of the response to treatment.
- Non-ferumoxytol Enhanced MRI: Patients scheduled for routine decompression surgery and autologous stem cell transplant receive follow-up magnetic resonance imaging in regular intervals for evaluation of the response to treatment.
Period: Overall Study
Arm/Group | Ferumoxytol-enhanced MRI | Non-ferumoxytol Enhanced MRI
Started | 9 | 5
Completed | 8 | 5
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ferumoxytol-enhanced MRI | Non-ferumoxytol Enhanced MRI | Total
Number analyzed (Participants) | 9 | 5 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 0 | 1
  Between 18 and 65 years | 8 | 5 | 13
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 5
  Male | 5 | 4 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 7 | 0 | 7
  Unknown or Not Reported | 1 | 5 | 6
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 9 | 5 | 14

OUTCOME MEASURES:

1. Primary Outcome: Signal to Noise Ratio (SNR)
Description: SNR is a measurement that compares the strength of a signal to the level of background noise. It is often expressed in decibels (dB) and is calculated by dividing the signal power by the noise power. A ratio greater than 1:1 indicates that there is more signal than noise.
  First, for each lesion the MR signal intensity (SI) of the lesion and the SI of the background (= noise in the image) was measured, then the SI of the lesion was divided by the SI of the noise to obtain the signal to noise ratio. Then, the mean SNR and standard deviation was calculated for the different groups of lesions and compared to the mean SNR between treated versus not treated lesions and treated lesions at different time points after the treatment using statistical tests.
Time Frame: week 1 postsurgery
Population: Participants who completed the protocol
Measure: Mean (Standard Deviation); unit: dB
Arm/Group | Ferumoxytol-enhanced MRI | Non-ferumoxytol Enhanced MRI
Number analyzed (Participants) | 8 | 5
dB | 33.82 (12.43) | 129.56 (10.93)
Statistical Analysis 1: Comparison: Ferumoxytol-enhanced MRI vs Non-ferumoxytol Enhanced MRI; Test type: Other; p = 0.002, Mixed Models Analysis — A p-value less than the a priori threshold of 0.05 was considered statistically significant; Mixed effects model including a random effect term accounting for correlation among the measures with a same patient

2. Primary Outcome: T2*-Relaxation Time
Description: T2* relaxation time is a measure of how quickly transverse magnetization decays in magnetic resonance imaging (MRI). It's a key factor in image contrast in gradient-echo (GRE) sequences and is used in many MRI applications, such as perfusion imaging, susceptibility-weighted imaging, and functional imaging. Lower T2* relaxation times indicate greater contrast agent uptake in cells.
Time Frame: week 1 postsurgery
Population: Participants who completed the protocol
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Ferumoxytol-enhanced MRI | Non-ferumoxytol Enhanced MRI
Number analyzed (Participants) | 8 | 5
milliseconds | 9.04 (0.7) | 13.7 (2.50)
Statistical Analysis 1: Comparison: Ferumoxytol-enhanced MRI vs Non-ferumoxytol Enhanced MRI; Test type: Other; p = 0.02, Mixed Models Analysis — A p-value less than the a priori threshold of 0.05 was considered statistically significant; Mixed effects model including a random effect term accounting for correlation among the measures with a same patient

3. Primary Outcome: Evaluation of Treatment Response to Decompression Surgery and Stem Cell Transplant
Description: Number of femurs that did not collapse by 1 year follow up. Evaluation of progression of osteonecrosis via scale 1-4, bone marrow edema, collapse of subchondral fractures.
Time Frame: one year
Population: Long-term follow up was conducted in the ferumoxytol group only
Measure: Count of Units; unit: Femur
Units Other Than Participants: Femur
Arm/Group | Ferumoxytol-enhanced MRI | Non-ferumoxytol Enhanced MRI
Number analyzed (Participants) | 8 | 0
Number analyzed (Femur) | 16 | 0
Femur | 12 |

ADVERSE EVENTS:
Time Frame: 1 week period (20 minute treatment and 1 week follow-up) plus follow-up visits for approximately 1 year
Arm/Group | Ferumoxytol-enhanced MRI | Non-ferumoxytol Enhanced MRI
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/5
Other Adverse Events (participants affected / at risk) | 0/9 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-04-11): https://cdn.clinicaltrials.gov/large-docs/93/NCT02893293/Prot_SAP_000.pdf
  • Informed Consent Form (2023-06-20): https://cdn.clinicaltrials.gov/large-docs/93/NCT02893293/ICF_001.pdf